CLINICAL TRIAL: NCT01986075
Title: A Sequenced Behavioral and Medication Intervention for Cocaine Dependence
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Frances R Levin, Director of Substance Use Disorder, New York State Psychiatric Institute
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #6850; R01DA034087-01A1 (NIH)
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Results first posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Cocaine Dependence
Keywords: Cocaine Dependence Treatment; Computer-assisted therapy; Pharmacotherapy
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — SLI381; TES

STUDY DESIGN:
Intervention Model Description: Following an initial 4 week period where participants received computer-assisted behavioral intervention based on the community reinforcement approach with contingency management (CRA + CM), individuals who failed to achieve abstinence will continue the behavioral treatment (CRA + CM) and will be randomly assigned, in parallel, to a behavioral therapy enhancement strategy that will include either Mixed Amphetamine Salts-Extended Release (80mg) or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Computer-assisted CBT plus Mixed-Amphetamine Salts- Extended Release (MAS-ER) (Experimental): Patients who are randomized to the computer-assisted behavior therapy plus mixed amphetamine salts (extended release) arm will have their dose titrated to 80 mg or the maximum tolerated extended release mixed amphetamine salts daily. Participants will be asked to take the medication once per day in the morning or early afternoon and will be maintained on this schedule through week 14 of the trial. Computer-assisted behavior therapy based on the Community Reinforcement Approach (CRA) to treating cocaine dependence. CRA is skills based treatment program that incorporates coping skills development and contingency management. Participants will attend the clinic 3x per week and receive counseling 2x per week.
  Interventions: Behavioral: Computer-assisted behavior therapy; Drug: Mixed-Amphetamine Salts- Extended Release (MAS-ER)
- Computer-assisted CBT plus placebo (Placebo Comparator): Patients who are randomized to the Computer-assisted CBT plus placebo arm will have their medication dose titrated in a fix-flexible dose schedule matching the active medication arm. Participants will be asked to take the medication once per day in the morning or early afternoon and will be maintained on this schedule through week 14 of the trial. Computer-assisted behavior therapy based on the Community Reinforcement Approach (CRA) to treating cocaine dependence. CRA is skills based treatment program that incorporates coping skills development and contingency management. Participants will attend the clinic 3x per week and receive counseling 2x per week.
  Interventions: Behavioral: Computer-assisted behavior therapy; Drug: Placebo

INTERVENTIONS:
Behavioral: Computer-assisted behavior therapy — TES is a computer-assisted therapy program delivered via effective informational and multimedia technologies, includes 32 core interactive, multimedia modules, beginning with basic cognitive behavioral relapse prevention skills (e.g. drug refusal skills) and moving on to improving psychosocial functioning, (e.g. employment status, social relations) and HIV risk reduction.
  Other Names: Therapeutic Educational System (TES)
Drug: Mixed-Amphetamine Salts- Extended Release (MAS-ER) — 80 mg/day of Mixed-Amphetamine Salts- Extended Release (MAS-ER) and computer -assisted CBT
  Other Names: Adderall XR
  Arms: Computer-assisted CBT plus Mixed-Amphetamine Salts- Extended Release (MAS-ER)
Drug: Placebo — Will receive computer -assisted CBT and placebo (instead of active Adderall-XR)
  Other Names: Computer-assisted CBT, TES
  Arms: Computer-assisted CBT plus placebo

SUMMARY:
This study will investigate a treatment strategy in which a computer-assisted behavioral intervention will be used to help individuals stop their use of cocaine. A medication will be combined with the behavioral treatment among those individuals who do not respond to the behavioral intervention alone. The primary hypothesis of the study is that among cocaine dependent individuals who fail to respond to an initial trial of behavioral therapy, a greater proportion of individuals will benefit from the combined treatment (behavior therapy plus medication) compared to individuals in the comparison group.

DETAILED DESCRIPTION:
Cocaine Dependence is associated with substantial social, physical, and neurobiological problems. Psychosocial treatments can be helpful for many individuals. However, a significant proportion of individuals do not benefit from counseling alone. Our research group has demonstrated that deficient dopamine transmission, predicts poor response to a behavioral treatment and that a regiment that included an agonist replacement strategy with stimulants maybe effective for promoting abstinence in severe cocaine dependent patients.

In this 15-week study 145 treatment-seeking cocaine dependent participants will receive a computer-assisted behavioral intervention based on the community reinforcement approach with contingency management (CRA + CM). The counseling approach will include both computer-assisted life skills training via and counseling. Individuals who fail to achieve abstinence will continue the behavioral treatment (CRA + CM) and will be randomly assigned to a behavioral therapy enhancement strategy that will include either Mixed Amphetamine Salts-Extended Release (80mg) or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Meets DSM-V criteria for cocaine use disorder.
2. Used cocaine at least four days in the past month.
3. Age 18-60.
4. Able to give informed consent and comply with study procedures

Exclusion Criteria:

1. Meets DSM-V criteria for bipolar disorder, schizophrenia or any psychotic disorder other than transient psychosis due to drug abuse.
2. Participants with MDD, with symptom severity that exceeds a HAM-D score of 20, and/or any other current Axis I psychiatric disorder as defined by DSM-V supported by the MINI that in the investigator's judgment are unstable, would be disrupted by study medication, or are likely to require specialized pharmacotherapy or psychotherapy during the study period.
3. History of seizures, unexplained loss of consciousness, or traumatic brain injury.
4. History of allergic reaction to candidate medication (amphetamine).
5. Significant current suicidal risk.
6. Pregnancy, lactation, or failure in sexually active female patients to use adequate contraceptive methods.
7. Unstable physical disorders which might make participation hazardous such as uncontrolled hypertension, acute hepatitis, uncontrolled diabetes.
8. Elevated transaminase levels (> 3x the normal limit).
9. Coronary vascular disease
10. History of failure to respond to a previous adequate trial of the candidate medication.
11. Current physiological dependence on any other substance other than nicotine or cannabis that would require a medically supervised detoxification.
12. Currently being prescribed psychotropic medication by another physician.
13. Are legally mandated (e.g. to avoid incarceration, monetary or other penalties, etc.) to participate in substance abuse treatment program.
14. Body Mass Index (BMI) < 18kg/m2. (amphetamine may produce weigh loss thus a minimum BMI cut-off is being used for study inclusion).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frances R Levin, M.D., Principal Investigator — Columbia University/New York State Psychiatric Institute
Locations (1):
- STARS, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bickel WK, Marsch LA, Buchhalter AR, Badger GJ. Computerized behavior therapy for opioid-dependent outpatients: a randomized controlled trial. Exp Clin Psychopharmacol. 2008 Apr;16(2):132-43. doi: 10.1037/1064-1297.16.2.132. PMID 18489017
- [Derived] Carpenter KM, Choi CJ, Basaraba C, Pavlicova M, Brooks DJ, Brezing CA, Bisaga A, Nunes EV, Mariani JJ, Levin FR. Mixed amphetamine salts-extended release (MAS-ER) as a behavioral treatment augmentation strategy for cocaine use disorder: A randomized clinical trial. Exp Clin Psychopharmacol. 2024 Feb;32(1):112-127. doi: 10.1037/pha0000676. Epub 2023 Sep 21. PMID 37732961
- [Derived] Blevins D, Carpenter KM, Martinez D, Mariani JJ, Levin FR. An adaptive clinical trial design for cocaine use disorder: Extended-release amphetamine salts for early behavioral intervention non-responders. Contemp Clin Trials. 2020 Nov;98:106187. doi: 10.1016/j.cct.2020.106187. Epub 2020 Oct 18. PMID 33086160
- See also: Click here for more information about the study and clinic — http://stars.columbia.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 145 participants enrolled, 21 participants were designated as treatment responders during the first month of the psychosocial intervention and were not randomized. An additional 38 individuals were lost to follow-up or not eligible to be randomized prior to completing the first month of the intervention. Eighty-six participants continued to use cocaine through the first month of treatment and were randomized to receive either MAS-XR or Placebo at the beginning of treatment week 5.
Groups:
- Computer-assisted CBT Plus Mixed-Amphetamine Salts- Extended Release (MAS-ER): Patients who are randomized to the computer-assisted behavior therapy plus mixed amphetamine salts (extended release) arm will have their dose titrated to 80 mg or the maximum tolerated extended release mixed amphetamine salts daily. Participants will be asked to take the medication once per day in the morning or early afternoon and will be maintained on this schedule through week 14 of the trial. Computer-assisted behavior therapy based on the Community Reinforcement Approach (CRA) to treating cocaine dependence. CRA is skills based treatment program that incorporates coping skills development and contingency management. Participants will attend the clinic 3x per week and receive counseling 2x per week.
  Computer-assisted behavior therapy: TES is a computer-assisted therapy program delivered via effective informational and multimedia technologies, includes 32 core interactive, multimedia modules, beginning with basic cognitive behavioral relapse prevention skills (e.g. drug refusal skills) and moving on to improving psychosocial functioning, (e.g. employment status, social relations) and HIV risk reduction.
  Mixed amphetamine salts: 80 mg/day of Mixed-Amphetamine Salts- Extended Release (MAS-ER) and computer -assisted CBT
- Computer- Assisted CBT With Contingency Management: All participants received computer-assisted CBT with contingency management (CRA + CM) during the first 4 week period of the trial.
Period: Initial CBT + CM (Pre-randomization)
Arm/Group | Computer-assisted CBT Plus Mixed-Amphetamine Salts- Extended Release (MAS-ER) | Computer-assisted CBT Plus Placebo | Computer- Assisted CBT With Contingency Management
Started | 0 | 0 | 145
Completed | 0 | 0 | 86
Not Completed | 0 | 0 | 59
Period: Randomized Intervention
Arm/Group | Computer-assisted CBT Plus Mixed-Amphetamine Salts- Extended Release (MAS-ER) | Computer-assisted CBT Plus Placebo | Computer- Assisted CBT With Contingency Management
Started | 45 | 41 | 0
Completed | 30 | 27 | 0
Not Completed | 15 | 14 | 0

BASELINE CHARACTERISTICS:
Groups:
- Non-randomized Individuals: Patients who were enrolled in the initial 4 week period and received CBT + CM but were not eligible to be randomized and did not enter the second randomized period of the trial.
- Total: Total of all reporting groups
Arm/Group | Computer-assisted CBT Plus Mixed-Amphetamine Salts- Extended Release (MAS-ER) | Computer-assisted CBT Plus Placebo | Non-randomized Individuals | Total
Number analyzed (Participants) | 45 | 41 | 59 | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (10.1) | 44.6 (9.8) | 42.9 (10.1) | 44.0 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 8 | 23
  Male | 38 | 33 | 51 | 122
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 9 | 15 | 35
  Not Hispanic or Latino | 34 | 32 | 44 | 110
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 3 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 20 | 17 | 23 | 60
  White | 19 | 20 | 22 | 61
  More than one race | 3 | 1 | 9 | 13
  Unknown or Not Reported | 2 | 0 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 45 | 41 | 59 | 145
Number of days of cocaine use during prior 28 days [Mean (Standard Deviation); unit: days] | 11.4 (6.1) | 13.9 (7.2) | 12.2 (7.4) | 12.6 (6.7)

OUTCOME MEASURES:

1. Primary Outcome: Those Achieving Three Consecutive Weeks of Cocaine Abstinence at the End of the Trial.
Description: The primary outcome measure will be a binary indicator (yes or no) of at least 3 consecutive weeks of urine toxicology confirmed self-reported abstinence during the last three weeks of the trial.
Time Frame: weeks 12-14 of trial
Measure: Count of Participants; unit: Participants
Arm/Group | Computer-assisted CBT Plus Mixed-Amphetamine Salts- Extended Release (MAS-ER) | Computer-assisted CBT Plus Placebo
Number analyzed (Participants) | 45 | 41
Participants | 7 | 5

ADVERSE EVENTS:
Time Frame: During 15 weeks of trial, or length of individual's participation
Description: Adverse events are reported for those individuals randomized to either of the two arms MAS-ER or placebo as well as those non-randomized individuals who received CBT plus CM
Groups:
- Computer-assisted CBT Plus Mixed-Amphetamine Salts- Extended Release (MAS-ER): Patients who are randomized to the computer-assisted behavior therapy plus mixed amphetamine salts (extended release) arm will have their dose titrated to 80 mg or the maximum tolerated extended release mixed amphetamine salts daily. Participants will be asked to take the medication once per day in the morning or early afternoon and will be maintained on this schedule through week 14 of the trial. Computer-assisted behavior therapy based on the Community Reinforcement Approach (CRA) to treating cocaine dependence. CRA is skills based treatment program that incorporates coping skills development and contingency management. Participants will attend the clinic 3x per week and receive counseling 2x per week.
  Computer-assisted behavior therapy: TES is a computer-assisted therapy program delivered via effective informational and multimedia technologies, includes 32 core interactive, multimedia modules, beginning with basic cognitive behavioral relapse prevention skills (e.g. drug refusal skills) and moving on to improving psychosocial functioning, (e.g. employment status, social relations) and HIV risk reduction.
  Mixed amphetamine salts: 80 mg/day of Adderall-XR and computer -assisted CBT
- Non-randomized CBT Plus CM: Fifty nine individuals who were not randomized and only exposed to CBT and CM. 21 participants were designated as treatment responders during the first month of the psychosocial intervention and were not randomized. An additional 38 individuals were lost to follow-up or not eligible to be randomized prior to completing the first month of the intervention.
Arm/Group | Computer-assisted CBT Plus Mixed-Amphetamine Salts- Extended Release (MAS-ER) | Computer-assisted CBT Plus Placebo | Non-randomized CBT Plus CM
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/41 | 0/59
Serious Adverse Events (participants affected / at risk) | 1/45 | 1/41 | 4/59
Other Adverse Events (participants affected / at risk) | 26/45 | 11/41 | 2/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Computer-assisted CBT Plus Mixed-Amphetamine Salts- Extended Release (MAS-ER) (N=45) | Computer-assisted CBT Plus Placebo (N=41) | Non-randomized CBT Plus CM (N=59)
inpatient rehabilitation stay (General disorders) | 0 (0) | 1 (1) | 1 (1)
dehydration (General disorders) | 1 (1) | 0 (0) | 0 (0)
hernia (General disorders) | 0 (0) | 0 (0) | 1 (1)
atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
GI issue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — participant swallowed a metal object
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Computer-assisted CBT Plus Mixed-Amphetamine Salts- Extended Release (MAS-ER) (N=45) | Computer-assisted CBT Plus Placebo (N=41) | Non-randomized CBT Plus CM (N=59)
insomnia (General disorders) | 14 (14) | 2 (2) | 0 (0)
anxiety (Psychiatric disorders) | 10 (10) | 3 (3) | 1 (1)
nausea (Gastrointestinal disorders) | 9 (9) | 2 (2) | 0 (0)
irritability (General disorders) | 5 (5) | 3 (3) | 0 (0)
hypertension (Cardiac disorders) | 6 (6) | 2 (2) | 0 (0)
headache (General disorders) | 3 (3) | 3 (3) | 1 (1)
appetite loss (General disorders) | 4 (4) | 1 (1) | 0 (0)
dry mouth (General disorders) | 4 (4) | 1 (1) | 0 (0)
constipation (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2013-10-31): https://cdn.clinicaltrials.gov/large-docs/75/NCT01986075/Prot_000.pdf
  • Statistical Analysis Plan (2012-07-05): https://cdn.clinicaltrials.gov/large-docs/75/NCT01986075/SAP_001.pdf